CLINICAL TRIAL: NCT00817674
Title: Sleep Disturbances as a Non-traditional Risk Factor in CKD-Wrist Actigraphy
Brief Title: Sleep Disturbances as a Non-traditional Risk Factor in CKD-Actigraphy
Acronym: CRIC
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: University of Illinois at Chicago (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Other Study IDs: #14081A; 5R01DK071696 (NIH)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Kidney Disease; Sleep Loss
Keywords: CKD; Kidney Disease; poor sleep; CKD progression
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: CKD subjects
- 2: Healthy Controls

SUMMARY:
To test if usual at home night time sleep duration as measured with activity monitors and questionnaires will predict changes in kidney function as measured by kidney filtration rate and of cardiovascular function as measured by C-reactive protein in the blood. The study will explore the role of decreased sleep time or decreased sleep quality as a non-traditional risk factor for the progression of CKD and for the development of cardiovascular disease in CKD.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate CKD
* Healthy controls age and gender matched to CKD subjects
* Regular bedtimes of at least 6h/night, sedentary lifestyle

Exclusion Criteria:

* Diabetes
* Current or previous dialysis for more than 1 month
* Uncontrolled hypertension
* Heart failure
* Liver disease
* HIV
* Hemoglobin < 10.5 g/dl
* Treatment with EProcrit, Epogen, or Aranesp
* Bone or organ transplant,
* Use of immunosuppressive drugs within past 6 months
* Current oral contraceptive use
* Current pregnancy
* Chemotherapy for malignancy within past 2 years

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD subjects; healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2007-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
CKD progression as measured by changes in GFR and cardiovascular risk as measured by CRP over a 5 year period | 5 years

SECONDARY OUTCOMES:
insulin resistance | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States